CLINICAL TRIAL: NCT04878159
Title: Association of Cardiac and Inflammatory Bio Markers and Morbidity in Emergency High-risk Abdominal Surgery
Brief Title: Troponin T and Emergency High-risk Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Sofia Kärnsund, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-21012302
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Emergency Laparotomy; Inflammatory Response; Myocardial Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency high-risk abdominal surgery: Patients undergoing emergency high-risk abdominal surgery, defined as immediate emergency laparoscopy or laparotomy, including intestinal obstruction, perforated viscus, intestinal ischemia and intraabdominal bleeding. Includes both primary surgery and re-operation after elective surgery.

SUMMARY:
To assess whether perioperatively elevated TnT levels, using high sensitivity troponin T (hsTnT) measurements, are associated with an increased risk of postoperative mortality as well as severe postoperative complications.

DETAILED DESCRIPTION:
Cardiac Troponin T (TnT) is a cardiac-specific molecule, released into the systemic circulation following myocardial cell injury. The release of cardiac Troponins is common during critical illness and is associated with increased morbidity and mortality. The mechanisms by which TnT is released in the blood during critical illness are not fully understood, but sepsis and inflammation are primary non-cardiac conditions during which elevated TnT levels are commonly seen. Previous research has shown that 84 percent of patients admitted to ICU had at least one elevated TnT measurement perioperatively. Patients undergoing high-risk abdominal surgery, defined as immediate emergency laparoscopy or laparotomy, are critically ill, often septic and with an acute inflammatory response and potential multiple organ system dysfunctions both prior but largely after surgery.

The hypothesis is that there is an association between elevated perioperative levels of cardiac Troponin T and mortality in patients undergoing emergency high-risk abdominal surgery.

The primary objective is to assess whether perioperatively elevated TnT levels, using high sensitivity troponin T (hsTnT) measurements, are associated with an increased risk of postoperative mortality as well as severe postoperative complications.

Patients requiring immediate emergency laparotomy or laparoscopy, including reoperations after elective gastrointestinal surgery and reoperations after previous non emergency high-risk abdominal surgery surgery, will be included in the study.

Two primary exposure measures will be investigated:

1. Peak Troponin T values ≥14 vs. Troponin T values <14. Patients with at least one measured Troponin T value ≥14 postoperatively will be allocated to the "elevated hsTnT" group
2. Postoperative hsTnT concentration ≥14 as well as a >50% relative increase from preoperative hsTnT concentration. Patients with hsTnT levels meeting these conditions will be allocated to the "elevated hsTnT" group hsTnT will be taken by blood samples preoperatively as well as on postoperative day 1, 2 and 3.

Primary analyses investigating the association between hsTnT and 30-day mortality (yes/no) and severe complications (yes/no) will be done using logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

Adults (18 years or over) undergoing emergency laparotomy or laparoscopy for following abdominal pathology:

* Intestinal obstruction
* Perforated viscus
* Intestinal ischemia
* Intraabdominal bleeding

The above conditions include both primary surgery and re-operation after elective surgery.

Exclusion Criteria:

Patients undergoing

* Appendicectomies
* Negative laparoscopies/laparotomies
* Cholecystectomies
* Simple herniotomies following incarceration without bowel resection
* Reoperation due to fascial separation with no other abdominal pathology identified
* Internal hernia after Roux-en-Y gastric bypass surgery
* Subacute surgery (surgery planned within 48 h) for inflammatory bowel diseases
* Subacute colorectal cancer surgery
* Patients with missing hsTnT values on both postoperative day 1 and 2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing emergency high-risk abdominal surgery at Hvidovre Hospital, Denmark, that meet the criteria for inclusion. Hvidovre hospital serves as the primary emergency hospital for more than 500 000 inhabitants.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days
Severe complication (Clavien Dindo ≥ 3) | 30 days

SECONDARY OUTCOMES:
Death | 90 days
Length of hospital stay | 30 days
Length of ICU stay | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No